CLINICAL TRIAL: NCT05121298
Title: Discontinuation of Methotrexate in Rheumatoid Arthritis Patients Achieving Clinical Remission by Treatment With Upadacitinib Plus Methotrexate: an Interventional, Multicenter, Prospective, Open-label, Single-arm Clinical Trial With Clinical, Ultrasound and Biomarker Assessments
Brief Title: Discontinuation of Methotrexate in Rheumatoid Arthritis Patients Achieving Clinical Remission by Treatment With Upadacitinib Plus Methotrexate
Acronym: DOPPLER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Atsushi Kawakami (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor-Investigator, Atsushi Kawakami, Professor, Nagasaki University
Organization: Nagasaki University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRB20-024
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Rheumatoid Arthritis; JAK Inhibitor; Musculoskeletal Ultrasound; Biomarker
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — upadacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Upadacitinib (Experimental): The administration of upadacitinib 15mg/day
  Interventions: Drug: upadacitinib 15mg/day

INTERVENTIONS:
Drug: upadacitinib 15mg/day — Patients will receive upadacitinib 15mg/day and continue to receive same doses of MTX until 24 weeks. If patients achieve a European League Against Rheumatism (EULAR) moderate response or a Disease Activity Score 28 (DAS28-CRP) ≤3.2 at 12 weeks, and a DAS28-CRP of <2.6 at 24 weeks, they will discontinue MTX, and continue upadacitinib until 48 weeks.

SUMMARY:
The administration of Janus kinase (JAK) inhibitors as well as biological disease-modifying anti-rheumatic drugs has dramatically improved even the clinical outcomes in rheumatoid arthritis (RA) patients with inadequate response to methotrexate (MTX). Upadacitinib is a selective JAK1 inhibitor to be approved for use in RA. Nearly half of patients added JAK inhibitors including upadacitinib can achieve clinical remission in RA patients with inadequate response to MTX. As the next step, it is the great issue whether disease activity can be maintained in good condition even if MTX is discontinued after achieving clinical remission in patients treated with the combination of JAK inhibitors and MTX. Thus, it is desirable to investigate the maintenance of clinical non-relapse after discontinuation of MTX in RA patients with clinical remission during treatment with upadacitinib plus MTX. In this study, we will evaluate the proportion of patients who maintained nonclinical relapse after discontinuation of MTX in patients with RA who achieved clinical remission after treatment with upadacitinib plus MTX. We will also use musculoskeletal ultrasound (MSUS) assessments to determine whether discontinuation of MTX can be maintained nonclinical relapse in RA patients achieving clinical remission.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following requirements to be considered for entry into the study:

  1. ≥20 years old
  2. with the diagnosis of RA based on the American College of Rheumatology (ACR) /EULAR 2010 RA Classification Criteria
  3. with at least moderate DAS28-CRP >3.2 at the eligibility evaluation
  4. with at least one PD score positive joint of 22 joints examined MSUS at the eligibility evaluation
  5. treated with MTX for ≥8 weeks prior to the providing consent, including 4 weeks or more at the same doses of 6 to 16 mg per week
  6. ability and willingness to provide written informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

* The exclusion criteria are as follows:

  (1) concurrent use of a corticosteroid equivalent to >7.5 mg/day of prednisolone (2) applicable an item for the contraindication of upadacitinib (3) a previous use of a JAK inhibitor (4) treatment with a corticosteroid and change of dose within 4 weeks prior to the providing consent (5) treatment with a csDMARD except MTX within 2 weeks prior to the providing consent; (6) treatment with a biologic DMARD or a biosimilar DMARD (ie, infliximab, biosimilar of infliximab, adalimumab, golimumab, certolizumab pegol, tocilizumab, sarilumab or abatacept) within 8 weeks prior to the providing consent (7) treatment with a TNF inhibitor (ie, etanercept or biosimilar of etanercept) within 4 weeks prior to the providing consent (8) use of a prohibited drug or therapy, other than the agents noted above, within 4 weeks prior to the providing consent (9) a complication causing musculoskeletal disorders other than RA (ie, ankylosing spondyloarthritis, reactive arthritis, psoriatic arthritis, crystal-induced arthritis, systemic lupus erythematosus, systemic scleroderma, inflammatory myopathy, or mixed connective tissue disease) (10) current pregnancy, breastfeeding, or noncompliant with a medically approved contraceptive regimen during and 12 months after the study period (11) inappropriateness for inclusion in this study as determined by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
maintenance of DAS28-CRP <=3.2 from week 24 to 48 in patients who achieve the DAS28-CRP <2.6 at week 24. | at week 48

SECONDARY OUTCOMES:
achievement of DAS28-CRP <=3.2 | at weeks 12, 24 and 36
achievement of DAS28-CRP <2.6 | at weeks 12, 24, 36 and 48
clinical relapse (DAS28-CRP >3.2) at week 48 in patients who achieve the DAS28-CRP <2.6 at week 24 | at week 48
achievement of EULAR moderate response | at week 12
changes in the DAS28-CRP value | from baseline to weeks 12, 24, 36, and 48
  Higher scores mean a more active RA.
changes in the DAS28-ESR value | from baseline to weeks 12, 24, 36, and 48
  Higher scores mean a more active RA.
changes in the DAS28-CRP value | from week 24 to weeks 36 and 48
  Higher scores mean a more active RA.
changes in the DAS28-ESR value | from week 24 to weeks 36 and 48
  Higher scores mean a more active RA.
changes in the clinical disease activity index (CDAI) value | from baseline to weeks 12, 24, 36, and 48
  Higher scores mean a more active of RA.
changes in the simplified disease activity index (SDAI) value | from baseline to weeks 12, 24, 36, and 48
  Higher scores mean a more active of RA.
changes in the clinical disease activity index (CDAI) value | from week 24 to weeks 36 and 48
  Higher scores mean a more active of RA.
changes in the simplified disease activity index (SDAI) value | from week 24 to weeks 36 and 48
  Higher scores mean a more active of RA.
achievement of CDAI <=2.8 | at weeks 12, 24, 36 and 48
achievement of SDAI <=3.3 | at weeks 12, 24, 36 and 48
changes in the serum levels of biomarkers | from baseline to weeks 12, 24, 36, and 48
  We analyze the serum levels of multiple biomarkers such as cytokines and chemokines.
changes in the serum levels of biomarkers | from week 24 to weeks 36 and 48
  We analyze the serum levels of multiple biomarkers such as cytokines and chemokines.
changes in the total power Doppler (PD) score | from baseline to weeks 12, 24, 36, and 48
  The minimum: 0, max: 66. Higher scores mean a more active RA.
changes in the total grayscale (GS) score | from baseline to weeks 12, 24, 36, and 48
  The minimum: 0, max: 66. Higher scores mean a more active RA.
changes in the combined PD score | from baseline to weeks 12, 24, 36, and 48
  The minimum: 0, max: 66. Higher scores mean a more active RA.
changes in the total PD score | from week 24 to weeks 36 and 48
  The minimum: 0, max: 66. Higher scores mean a more active RA.
changes in the total GS score | from week 24 to weeks 36 and 48
  The minimum: 0, max: 66. Higher scores mean a more active RA.
changes in the combined PD score | from week 24 to weeks 36 and 48
  The minimum: 0, max: 66. Higher scores mean a more active RA.
change in van der Heijde-modified total Sharp score (vdH-mTSS) | from baseline to weeks 12, 24, 36 and 48
  The minimum: 0, max: 3. Higher scores mean a more joint destruction and deformity.
change in vdH-mTSS | from week 24 to weeks 36 and 48
  Higher scores mean a more joint destruction and deformity.

CONTACTS AND LOCATIONS:
Overall Officials: Atsushi Kawakami, MD, PhD, Principal Investigator — Nagasaki University
Locations (1):
- Nagasaki University Hospital, Nagasaki, Japan

REFERENCES:
- [Derived] Shimizu T, Kawashiri SY, Sato S, Kawazoe Y, Kuroda S, Kawasaki R, Ito Y, Morimoto S, Yamamoto H, Kawakami A. Discontinuation of methotrexate in rheumatoid arthritis patients achieving clinical remission by treatment with upadacitinib plus methotrexate (DOPPLER study): A study protocol for an interventional, multicenter, open-label and single-arm clinical trial with clinical, ultrasound and biomarker assessments. Medicine (Baltimore). 2022 Jan 14;101(2):e28463. doi: 10.1097/MD.0000000000028463. PMID 35029189